CLINICAL TRIAL: NCT06397781
Title: Effect of S. Aureus Skin Decolonization on Disease Severity in Atopic Dermatitis Patients
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Wanda Phipatanakul, S. Jean Emans, MD Professor of Pediatrics, Harvard Medical School (HMS and HSDM)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-P00047752
Record Dates: First submitted 2024-04-30; First posted 2024-05-03 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Skin Cleansing Regimen (Experimental): 1. Mupirocin 2% nasal ointment to the anterior nares to be applied twice daily
  2. Chlorhexidine 4% topical soap (Hibiclens) to be used every other day in the shower or bath from the neck down and then completely rinsed.
  3. Sulfamethoxazole/trimethoprim (Bactrim): one double strength (DS) tablet (800 mg/160 mg) twice per day for adolescents and adults
  Interventions: Drug: Skin Cleanser Combination No.1

INTERVENTIONS:
Drug: Skin Cleanser Combination No.1 — 1. Mupirocin 2% nasal ointment to the anterior nares to be applied twice daily
  2. Chlorhexidine 4% topical soap (Hibiclens) to be used every other day in the shower or bath from the neck down and then completely rinsed.
  3. Sulfamethoxazole/trimethoprim (Bactrim): one double strength (DS) tablet (800 mg/160 mg) twice per day for adolescents and adults. Dosing for pediatric patients will be calculated to 5 to 6 mg/kg trimethoprim also given twice daily.

SUMMARY:
Our hypothesis is that S. aureus skin decolonization in atopic dermatitis reduces disease severity and favorably alters the function and gene expression of epidermal and immune skin cells that contribute to disease severity.

DETAILED DESCRIPTION:
Patients will sign an informed consent and assent to participate. Skin and both nares will be cultured for S aureus. A blood sample and two 2 mm skin biopsies will be obtained one from non-lesional skin and another one from lesional skin). The patients will be instructed in the use of the three-week S. aureus decolonization regimen and provided with the medications (sulfamethoxazole/trimethoprim and Mupirocin ointment) and Chlorhexidine. The second visit will take place immediately at the end of the three-week S. aureus skin decolonization regimen. Disease severity will be assessed, the skin and nares will be re-cultured, and skin biopsies and blood will be obtained.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants ≥6 yrs of age
2. Meet atopic dermatitis Standard Diagnostic Criteria
3. SCORAD > 40.

Exclusion Criteria:

1. . Enrollment in another clinical trial
2. Hypersensitivity to an agent used for the skin decolonization protocol
3. Use within 4 weeks of systemic treatment with immunosuppressive/immunomodulating drugs (corticosteroids, cyclosporine, mycophenolate, azathioprine, methotrexate)
4. Phototherapy for AD within 4 weeks
5. Treatment with biologics (dupilumab, omalizumab, benralizumab, etc) within sixteen weeks
6. Use of topical steroids, topical calcineurin inhibitors within 7 days
7. Bleach baths within 7 days of the first Visit
8. Use of oral or topical antibiotics within 21 days of the beginning of the study
9. Asthmatics receiving more than 500 μg per day of inhaled corticosteroids
10. History of (HIV, hepatitis B, hepatitis C, tuberculosis malignancy
11. Skin comorbidities that may interfere with assessments: psoriasis, cutaneous T Cell lymphoma,,
12. Severe ongoing medical illnesses e.g. cardiovascular, renal disease, autoimmune disease.
13. Febrile illness at time of visits
14. Suspected immune deficiency or family history of primary immunodeficiency
15. Pregnancy

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2031-01-01 (Estimated); Primary Completion 2035-12 (Estimated); Study Completion 2039-12 (Estimated)

PRIMARY OUTCOMES:
Severity Scoring of Atopic Dermatitis Index | 3 weeks
  severity index

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States